CLINICAL TRIAL: NCT07063693
Title: Phase 1 Trial of ABY-029 Fluorescence in Patients With High-Grade Glioma
Brief Title: ABY-029 Glioma Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Linton T. Evans, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02002497; R01CA167413 (NIH)
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Intracranial Tumor
Keywords: ABY-029; Affibody; Molecular Fluorescence-Guided Surgery; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Brain Neoplasms | interventions — ABY-029

STUDY DESIGN:
Intervention Model Description: Sixteen participants with EGFR-positive tumors will be enrolled, alternating between two ABY-029 administration doses (the 6X dose and 10X dose), until eight participants with EGFR-positive tumors have been enrolled at each dose group. Because some participants may have EGFR-negative tumors, it may be necessary to enroll up to 33 participants before the target enrollment (eight participants with EGFR-positive tumors at each of two ABY-029 doses) is met.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABY-029 6X dose group (Experimental): ABY-029 will be administered at the 6X dose level prior to surgery to participants with presumed high-grade glioma, based on a preoperative MRI or other imaging. Investigators will collect one blood sample before participants are given ABY-029, a second sample one or two minutes after participants are given the drug, a third sample about 15 minutes after participants are given the drug, and a fourth sample about an hour after receiving the drug, or just prior to anesthesia (whichever comes first). Investigators will collect one urine sample and take EKG readings to monitor the participant's heart before surgery. Investigators will repeat blood, urine and EKG tests when participants are in the hospital after surgery.
  Interventions: Drug: ABY-029
- ABY-029 10X dose group (Experimental): ABY-029 will be administered at the 10X dose level prior to surgery to participants with presumed high-grade glioma, based on a preoperative MRI or other imaging. Investigators will collect one blood sample before participants are given ABY-029, a second sample one or two minutes after participants are given the drug, a third sample about 15 minutes after participants are given the drug, and a fourth sample about an hour after receiving the drug, or just prior to anesthesia (whichever comes first). Investigators will collect one urine sample and take EKG readings to monitor the participant's heart before surgery. Investigators will repeat blood, urine and EKG tests when participants are in the hospital after surgery.
  Interventions: Drug: ABY-029

INTERVENTIONS:
Drug: ABY-029 — ABY-029 will be administered via single intravenous injection to subjects with high-grade glioma approximately 1-3 hours prior to surgery.
  All research procedures will occur during surgery. The research procedures involve image and measurement data collection and biopsy specimen sampling. Research data collection will occur at 3 or 4 time points during surgery using either standard-of-care tools and methods or non-significant risk experimental devices.
  No follow-up visit will be required of participants. Participants will be monitored for possible adverse events for approximately 30 days by the operating surgeon involved in the clinical trial procedures and through review of participant medical records.

SUMMARY:
The purposes of the research trial are to study the safety of ABY-029 and to understand how much of the drug is needed to reach brain tumors so it can be visualized best by surgeons. Investigators will do this by comparing two groups of participants that receive different, very small amounts of ABY-029. Investigators will use an imaging system during surgery to record the amount of ABY-029 in the participant's tumor and in the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of presumed high-grade glioma, based on image data.
2. Tumor judged to be suitable and planned for open cranial resection.
3. Valid informed consent by participant.
4. Age ≥ 18 years old.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prisoners
2. Individuals who are pregnant or breast feeding.
3. Participants on any experimental or approved anti-EGFR targeted therapies
4. Elevated kidney or liver function tests (levels greater than 2.5 times the normal limit) from laboratory tests conducted as part of standard-of-care screening of prospective surgical participants no earlier than 30 days prior to surgery.
5. Any condition which, in the opinion of the clinical investigator, contraindicates research participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to ABY-029 | One month
  To study the safety of ABY-029, adverse events related to 6X and 10X doses of ABY-029 will be tracked following surgery, and the proportion of study-drug related adverse events at 6X and 10X doses will be compared statistically for significant differences.
False negative rate of ABY-029 fluorescence | Up to three months
  To measure of diagnostic performance of ABY-029, the false negative rate of ABY-029 fluorescence measured during surgery in tissue samples that are confirmed to be tumor through pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Linton Evans, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: No